CLINICAL TRIAL: NCT00105287
Title: Multi-center Study Evaluating OraVescent Fentanyl Citrate for the Treatment of Breakthrough Pain in Opioid Tolerant Cancer Patients
Brief Title: Treatment of Breakthrough Pain in Opioid Tolerant Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25608/3039/BP/US
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Pain; Cancer
Keywords: cancer; pain; Breakthrough Pain in cancer patients
MeSH Terms: conditions — Pain; Neoplasms

INTERVENTIONS:
Drug: OraVescent fentanyl (OVF)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of OraVescent fentanyl when used long-term to relieve breakthrough pain in opioid tolerant cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of a malignant solid tumor or hematological malignancy causing cancer related pain
* Currently taking around the clock opioid therapy for pain
* Experience on average, 1-4 breakthrough pain episodes per day

Exclusion Criteria:

* Opioid or fentanyl intolerance
* Sleep apnea or active brain metastases with increased intracranial pressure
* COPD (chronic obstructive pulmonary disease); cardiopulmonary disease; heart disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Primary Completion 2006-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Cullman Oncology and Hematology, Cullman, Alabama
  - Advanced Clinical Research Institute, Anaheim, California
  - Pacific Cancer Medical Center, Anaheim, California
  - Compassionate Cancer Care Medical Group, Corona, California
  - Compassionate Cancer Center, Fountain Valley, California
  - Clinical Trials & Research Associates, Inc., Montebello, California
  - San Diego Hospice & Palliative Care, San Diego, California
  - Pacific Clinical Research, Santa Monica, California
  - Lovelace Scientific Resources, Miami, Florida
  - Gulf Coast Pain Specialists, Pensacola, Florida
  - Hematology Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Center for Prospective Outcome, Marietta, Georgia
  - Iowa Pain Management Clinic, PC, Des Moines, Iowa
  - Donald Berdeaux, Great Falls, Montana
  - Great Falls Clinic, LLP, Great Falls, Montana
  - Southern Nevada Cancer Research, Las Vegas, Nevada
  - NYU Pain Management Center, New York, New York
  - Research Across America, New York, New York
  - Brody School of Medicine, Greenville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Charleston Hematology Oncology, PA, Charleston, South Carolina
  - University of Rochester, San Antonio, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Cache Valley Cancer Treatment and Research Clinic, Inc., West Point, Utah